CLINICAL TRIAL: NCT04729309
Title: Open-Label Study to Investigate the Mass Balance and Absolute Bioavailability of a Single Oral Dose of [14C]-Labeled RO7049389 or RO7049389 and an Intravenous Micro-Dose of [13C]-Labeled RO7049389 in Healthy Volunteers
Brief Title: Mass Balance and Absolute Bioavailability Study of RO7049389 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BP41811
Record Dates: First submitted 2021-01-26; First posted 2021-01-28 (Actual); Results first posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mass Balance (MB) Cohort (Experimental): Participants will receive oral [14C] RO7049389 under fasted conditions, followed by intravenous IV [13C] after a two-hour period.
  Interventions: Drug: [13C] RO7049389; Drug: [14C] RO7049389
- Absolute Bioavailability (BA) Cohort (Experimental): In Periods 1 and 2, participants will receive oral [12C] RO7049389 under fasted conditions, followed by IV [13C] RO7049389. There is a minimum 7-day washout between periods.
  Interventions: Drug: [12C] RO7049389; Drug: [13C] RO7049389

INTERVENTIONS:
Drug: [12C] RO7049389 — Participants will receive oral [12C] RO7049389.
  Arms: Absolute Bioavailability (BA) Cohort
Drug: [13C] RO7049389 — Participants will receive IV [13C] RO7049389.
Drug: [14C] RO7049389 — Participants will receive an oral suspension of [14C] RO7049389.
  Arms: Mass Balance (MB) Cohort

SUMMARY:
The objective of this study is to characterize the mass balance, absolute bioavailability, route and rates of elimination of RO7049839.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian (must have Caucasian parents and grandparents) or East Asian (must have Chinese, Korean, or Japanese parents and grandparents)
* Body mass index between 18 to 30 kg/m^2 (inclusive) and a weight range of 50 kg to 100 kg (inclusive) at screening
* For women of childbearing potential: agree to use two methods of contraception, with at least one method considered as highly effective during the study and for at least 90 days after the last dose of study drug
* For men: agree to remain abstinent (refrain from heterosexual intercourse) or agree to use contraceptive measures, and agree to refrain from donating sperm during the treatment period and for at least 90 days after the last dose of study drug

Exclusion Criteria:

* Pregnant or lactating women, and male participants with partners who are pregnant or lactating
* History or symptoms of any clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, oncologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study treatment; or of interfering with the interpretation of data
* Personal history or family history of congenital long QT interval (QT) syndrome and/or cardiac sudden death
* History of Gilbert syndrome
* Participants who have had significant acute infection, e.g. influenza, local infection, acute gastrointestinal (GI) symptoms, or any other clinically significant illness within two weeks of dose administration
* Any confirmed significant reactions (urticaria or anaphylaxis) against any drug, or multiple drug allergies
* Any clinically significant concomitant diseases or conditions that could interfere with the conduct of the study, or in the opinion of the Investigator, would pose an unacceptable risk to the participant in this study
* Taking any herbal medications or substances, supplements (including vitamins), traditional Chinese medicines, prescription medicine, or over-the-counter medications within 14 days of first dosing or within 5 times the elimination half-life of the medication prior to first dosing, whichever is longer
* History of having received any systemic anti-neoplastic (including radiation) or immune-modulatory treatment (including systemic oral or inhaled corticosteroids) 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
* Are currently enrolled in or have participated in any other clinical study involving an investigational product or in any other type of medical research within the last 90 days (or within 5 half-lives of the investigational product, whichever is longer)
* Donation or loss of blood or blood products in excess of 500 mL within 3 months of screening
* Evidence of current severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection
* Hepatitis A, B, C, D, or E or HIV infection
* History of drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in males > 21 units per week and in females > 14 units per week (1 unit = 1/2 pint of beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type)
* Use of > 5 cigarettes or equivalent nicotine-containing product per day prior to screening

Exclusion Criteria for Mass Balance Cohorts

* Regular work with ionizing radiation or radioactive material
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton [excluding spinal column]), during work, or during participation in a medical trial in the previous year
* History of gastrointestinal (GI) surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- Absolute Bioavailability (BA) Cohort: Period 1: Participants received 600 mg of oral [12C] RO7049389 under fasted conditions, followed by 100 ug of intravenous (IV) [13C] RO7049389 after a two-hour delay.
  Period 2: After a 7-day washout period, participants received 1000 mg of oral [12C] RO7049389, followed by 100 ug of IV [13C] RO7049389 after a two-hour delay.
- Mass Balance (MB) Cohort: Participants received 600 mg of [14C] RO7049389 oral suspension under fasted conditions, followed by 100 ug of intravenous (IV) [13C] RO7049389 after a two-hour delay. (Note: [14C] RO7049389 was a combination of [12C]+[14C]-labeled RO7049389).
Period: Period 1
Arm/Group | Absolute Bioavailability (BA) Cohort | Mass Balance (MB) Cohort
Started | 16 | 6
Completed | 12 | 6
Not Completed | 4 | 0
Not completed — Subject unable to return for Period 2 | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Period 2
Arm/Group | Absolute Bioavailability (BA) Cohort | Mass Balance (MB) Cohort
Started | 12 | 0
Completed | 12 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Absolute Bioavailability (BA) Cohort | Mass Balance (MB) Cohort | Total
Number analyzed (Participants) | 16 | 6 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 6 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (5.9) | 50.5 (7.7) | 35.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 9
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Dose Excreted in Urine - MB Cohort
Time Frame: Up to Day 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Mass Balance (MB) Cohort
Number analyzed (Participants) | 6
Percentage | 3.81 (35.2)

2. Primary Outcome: Percentage of Dose Excreted in Feces - MB Cohort
Time Frame: Up to Day 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Mass Balance (MB) Cohort
Number analyzed (Participants) | 6
Percentage | 90.5 (4.9)

3. Primary Outcome: Percent Total Recovery (Urine + Feces) - MB Cohort
Time Frame: Up to Day 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Mass Balance (MB) Cohort
Number analyzed (Participants) | 6
Percentage | 94.5 (5.5)

4. Primary Outcome: Absolute Oral BA for RO7049389 - BA Cohort
Time Frame: Up to Day 4 of Periods 1 and 2
Population: All participants who have received at least one dose of study treatment and who have data from at least one post-dose sample were included in the PK analysis population. Participants were excluded from the PK analysis population if they significantly violated the inclusion or exclusion criteria, deviated significantly from the protocol, or if data were unavailable or incomplete which may influence the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Absolute Bioavailability (BA) Cohort
Number analyzed (Participants) | 16
Percentage
  Asian participants - Period 1: number analyzed (Participants) | 8
  Asian participants - Period 1 | 41.7 (65.3)
  Caucasian participants - Period 1: number analyzed (Participants) | 7
  Caucasian participants - Period 1 | 30.6 (45.8)
  Asian participants - Period 2: number analyzed (Participants) | 5
  Asian participants - Period 2 | 61.4 (90.2)
  Caucasian participants - Period 2: number analyzed (Participants) | 5
  Caucasian participants - Period 2 | 40.7 (56)

5. Secondary Outcome: Clearance (CL) of RO7049389 - MB Cohort
Time Frame: Up to Day 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Mass Balance (MB) Cohort
Number analyzed (Participants) | 6
L/h
  [12C] RO7049389 | 100 (71.4)
  [13C] RO7049389 | 25.3 (54.3)

6. Secondary Outcome: Clearance (CL) of RO7049389 - BA Cohort
Time Frame: Up to Day 4 of Periods 1 and 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Absolute Bioavailability (BA) Cohort
Number analyzed (Participants) | 16
L/h
  Asian participants - [12C] Period 1: number analyzed (Participants) | 8
  Asian participants - [12C] Period 1 | 36.6 (122.3)
  Caucasian participants - [12C] Period 1: number analyzed (Participants) | 7
  Caucasian participants - [12C] Period 1 | 75.3 (69.2)
  Asian participants - [13C] Period 1: number analyzed (Participants) | 7
  Asian participants - [13C] Period 1 | 14.8 (48.2)
  Caucasian participants - [13C] Period 1: number analyzed (Participants) | 7
  Caucasian participants - [13C] Period 1 | 21.9 (28.7)
  Asian participants - [12C] Period 2: number analyzed (Participants) | 5
  Asian participants - [12C] Period 2 | 37.2 (152.1)
  Caucasian participants - [12C] Period 2: number analyzed (Participants) | 6
  Caucasian participants - [12C] Period 2 | 87.3 (96.5)
  Asian participants - [13C] Period 2: number analyzed (Participants) | 4
  Asian participants - [13C] Period 2 | 14.7 (43.9)
  Caucasian participants - [13C] Period 2: number analyzed (Participants) | 4
  Caucasian participants - [13C] Period 2 | 24.7 (42.3)

7. Secondary Outcome: Half-Life (T1/2) of RO7049389 - MB Cohort
Time Frame: Up to Day 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Mass Balance (MB) Cohort
Number analyzed (Participants) | 6
Hours
  [12C] RO7049389 | 8.1 (24.6)
  [13C] RO7049389 | 1.9 (23.6)
  [14C] RO7049389 | 11.4 (35.3)

8. Secondary Outcome: Half-Life (T1/2) of RO7049389 - BA Cohort
Time Frame: Up to Day 4 of Periods 1 and 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Absolute Bioavailability (BA) Cohort
Number analyzed (Participants) | 16
Hours
  Asian participants - [12C] Period 1: number analyzed (Participants) | 8
  Asian participants - [12C] Period 1 | 8.3 (35.4)
  Caucasian participants - [12C] Period 1: number analyzed (Participants) | 7
  Caucasian participants - [12C] Period 1 | 7.6 (31.1)
  Asian participants - [13C] Period 1: number analyzed (Participants) | 7
  Asian participants - [13C] Period 1 | 1.6 (32.8)
  Caucasian participants - [13C] Period 1: number analyzed (Participants) | 7
  Caucasian participants - [13C] Period 1 | 1.3 (46.0)
  Asian participants - [12C] Period 2: number analyzed (Participants) | 5
  Asian participants - [12C] Period 2 | 6.7 (83.6)
  Caucasian participants - [12C] Period 2: number analyzed (Participants) | 6
  Caucasian participants - [12C] Period 2 | 11.1 (34.6)
  Asian participants - [13C] Period 2: number analyzed (Participants) | 4
  Asian participants - [13C] Period 2 | 1.6 (36.7)
  Caucasian participants - [13C] Period 2: number analyzed (Participants) | 4
  Caucasian participants - [13C] Period 2 | 1.1 (46.7)

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of RO7049389 - MB Cohort
Time Frame: Up to Day 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Mass Balance (MB) Cohort
Number analyzed (Participants) | 6
ng/mL
  [12C] RO7049389 | 3820 (144.8)
  [13C] RO7049389 | 7.6 (16.9)
  [14C] RO7049389 | 6390 (89.7)

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) of RO7049389 - BA Cohort
Time Frame: Up to Day 4 of Periods 1 and 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Absolute Bioavailability (BA) Cohort
Number analyzed (Participants) | 16
ng/mL
  Asian participants - [12C] Period 1: number analyzed (Participants) | 8
  Asian participants - [12C] Period 1 | 6390 (118)
  Caucasian participants - [12C] Period 1: number analyzed (Participants) | 8
  Caucasian participants - [12C] Period 1 | 3000 (112.9)
  Asian participants - [13C] Period 1: number analyzed (Participants) | 8
  Asian participants - [13C] Period 1 | 8.2 (21.4)
  Caucasian participants - [13C] Period 1: number analyzed (Participants) | 8
  Caucasian participants - [13C] Period 1 | 7.7 (13.5)
  Asian participants - [12C] Period 2: number analyzed (Participants) | 5
  Asian participants - [12C] Period 2 | 9470 (110.7)
  Caucasian participants - [12C] Period 2: number analyzed (Participants) | 7
  Caucasian participants - [12C] Period 2 | 3570 (109.3)
  Asian participants - [13C] Period 2: number analyzed (Participants) | 5
  Asian participants - [13C] Period 2 | 8.7 (13.3)
  Caucasian participants - [13C] Period 2: number analyzed (Participants) | 6
  Caucasian participants - [13C] Period 2 | 7.7 (14.1)

11. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of RO7049389 - MB Cohort
Time Frame: Up to Day 17
Measure: Median (Full Range); unit: Hours
Arm/Group | Mass Balance (MB) Cohort
Number analyzed (Participants) | 6
Hours
  [12C] RO7049389 | 1.50 [1.00 to 2.00]
  [13C] RO7049389 | 2.13 [2.13 to 2.13]
  [14C] RO7049389 | 4.00 [1.50 to 8.00]

12. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of RO7049389 - BA Cohort
Time Frame: Up to Day 4 of Periods 1 and 2
Population: as for outcome 4
Measure: Median (Full Range); unit: Hours
Arm/Group | Absolute Bioavailability (BA) Cohort
Number analyzed (Participants) | 16
Hours
  Asian participants - [12C] Period 1: number analyzed (Participants) | 8
  Asian participants - [12C] Period 1 | 1.75 [1.50 to 2.00]
  Caucasian participants - [12C] Period 1: number analyzed (Participants) | 8
  Caucasian participants - [12C] Period 1 | 2.00 [1.00 to 4.00]
  Asian participants - [13C] Period 1: number analyzed (Participants) | 8
  Asian participants - [13C] Period 1 | 2.13 [2.13 to 2.13]
  Caucasian participants - [13C] Period 1: number analyzed (Participants) | 8
  Caucasian participants - [13C] Period 1 | 6.00 [4.00 to 8.00]
  Asian participants - [12C] Period 2: number analyzed (Participants) | 5
  Asian participants - [12C] Period 2 | 1.50 [1.50 to 2.00]
  Caucasian participants - [12C] Period 2: number analyzed (Participants) | 7
  Caucasian participants - [12C] Period 2 | 2.00 [1.00 to 4.00]
  Asian participants - [13C] Period 2: number analyzed (Participants) | 5
  Asian participants - [13C] Period 2 | 2.13 [2.13 to 2.13]
  Caucasian participants - [13C] Period 2: number analyzed (Participants) | 6
  Caucasian participants - [13C] Period 2 | 2.13 [2.13 to 2.13]

13. Secondary Outcome: Area Under Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of RO7049389 - MB Cohort
Time Frame: Up to Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Mass Balance (MB) Cohort
Number analyzed (Participants) | 6
h*ng/mL
  [12C] RO7049389 | 5970 (71.4)
  [13C] RO7049389 | 4.0 (54.3)
  [14C] RO7049389 | 83700 (39.6)

14. Secondary Outcome: Area Under Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of RO7049389 - BA Cohort
Time Frame: Up to Day 4 of Periods 1 and 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Absolute Bioavailability (BA) Cohort
Number analyzed (Participants) | 16
h*ng/mL
  Asian participants - [12C] Period 1: number analyzed (Participants) | 8
  Asian participants - [12C] Period 1 | 16400 (122.3)
  Caucasian participants - [12C] Period 1: number analyzed (Participants) | 7
  Caucasian participants - [12C] Period 1 | 7970 (69.2)
  Asian participants - [13C] Period 1: number analyzed (Participants) | 7
  Asian participants - [13C] Period 1 | 6.8 (48.2)
  Caucasian participants - [13C] Period 1: number analyzed (Participants) | 7
  Caucasian participants - [13C] Period 1 | 4.6 (28.7)
  Asian participants - [12C] Period 2: number analyzed (Participants) | 5
  Asian participants - [12C] Period 2 | 26900 (152.1)
  Caucasian participants - [12C] Period 2: number analyzed (Participants) | 6
  Caucasian participants - [12C] Period 2 | 11500 (96.5)
  Asian participants - [13C] Period 2: number analyzed (Participants) | 4
  Asian participants - [13C] Period 2 | 6.8 (43.9)
  Caucasian participants - [13C] Period 2: number analyzed (Participants) | 4
  Caucasian participants - [13C] Period 2 | 4.1 (42.3)

15. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUClast) of RO7049389 - MB Cohort
Time Frame: Up to Day 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Mass Balance (MB) Cohort
Number analyzed (Participants) | 6
h*ng/mL | 8280 (129.7)

16. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUClast) of RO7049389 - BA Cohort
Time Frame: Up to Day 4 of Periods 1 and 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Absolute Bioavailability (BA) Cohort
Number analyzed (Participants) | 16
h*ng/mL
  Asian participants - [12C] Period 1: number analyzed (Participants) | 8
  Asian participants - [12C] Period 1 | 16300 (123.1)
  Caucasian participants - [12C] Period 1: number analyzed (Participants) | 8
  Caucasian participants - [12C] Period 1 | 8110 (63.7)
  Asian participants - [13C] Period 1: number analyzed (Participants) | 8
  Asian participants - [13C] Period 1 | 6.5 (45.9)
  Caucasian participants - [13C] Period 1: number analyzed (Participants) | 8
  Caucasian participants - [13C] Period 1 | 4.4 (27.2)
  Asian participants - [12C] Period 2: number analyzed (Participants) | 5
  Asian participants - [12C] Period 2 | 26800 (152.2)
  Caucasian participants - [12C] Period 2: number analyzed (Participants) | 7
  Caucasian participants - [12C] Period 2 | 10100 (96.9)
  Asian participants - [13C] Period 2: number analyzed (Participants) | 5
  Asian participants - [13C] Period 2 | 7.2 (41.1)
  Caucasian participants - [13C] Period 2: number analyzed (Participants) | 6
  Caucasian participants - [13C] Period 2 | 4.3 (38.1)

17. Secondary Outcome: Apparent Clearance (CL/F) of RO7049389 - MB Cohort
Time Frame: Up to Day 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Mass Balance (MB) Cohort
Number analyzed (Participants) | 6
L/h | 100 (71.4)

18. Secondary Outcome: Apparent Clearance (CL/F) of RO7049389 - BA Cohort
Time Frame: Up to Day 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Absolute Bioavailability (BA) Cohort
Number analyzed (Participants) | 16
L/h
  Asian participants - [12C] Period 1: number analyzed (Participants) | 8
  Asian participants - [12C] Period 1 | 36.6 (122.3)
  Caucasian participants - [12C] Period 1: number analyzed (Participants) | 7
  Caucasian participants - [12C] Period 1 | 75.3 (69.2)
  Asian participants - [12C] Period 2: number analyzed (Participants) | 5
  Asian participants - [12C] Period 2 | 37.2 (152.1)
  Caucasian participants - [12C] Period 2: number analyzed (Participants) | 6
  Caucasian participants - [12C] Period 2 | 87.3 (96.5)
  Asian participants - [13C] Period 1: number analyzed (Participants) | 7
  Asian participants - [13C] Period 1 | 14.8 (48.2)
  Caucasian participants - [13C] Period 1: number analyzed (Participants) | 7
  Caucasian participants - [13C] Period 1 | 21.9 (28.7)
  Asian participants - [13C] Period 2: number analyzed (Participants) | 4
  Asian participants - [13C] Period 2 | 14.7 (43.9)
  Caucasian participants - [13C] Period 2: number analyzed (Participants) | 4
  Caucasian participants - [13C] Period 2 | 24.7 (42.3)

19. Secondary Outcome: Renal Clearance (CLr) of RO7049389 - BA Cohort
Time Frame: Up to Day 4 of Periods 1 and 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Absolute Bioavailability (BA) Cohort
Number analyzed (Participants) | 16
mL/min
  Asian participants - [12C] Period 1: number analyzed (Participants) | 8
  Asian participants - [12C] Period 1 | 2.7 (42.6)
  Caucasian participants - [12C] Period 1: number analyzed (Participants) | 8
  Caucasian participants - [12C] Period 1 | 1.1 (61.1)
  Asian participants - [12C] Period 2: number analyzed (Participants) | 5
  Asian participants - [12C] Period 2 | 2.5 (22.9)
  Caucasian participants - [12C] Period 2: number analyzed (Participants) | 7
  Caucasian participants - [12C] Period 2 | 0.8 (65.5)

20. Secondary Outcome: Amount Excreted in Urine (Ae) of RO7049389 - BA Cohort
Time Frame: Up to Day 4 of Periods 1 and 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Absolute Bioavailability (BA) Cohort
Number analyzed (Participants) | 16
mg
  Asian participants - [12C] Period 1: number analyzed (Participants) | 8
  Asian participants - [12C] Period 1 | 3.4 (2.5)
  Caucasian participants - [12C] Period 1: number analyzed (Participants) | 8
  Caucasian participants - [12C] Period 1 | 0.8 (0.8)
  Asian participants - [12C] Period 2: number analyzed (Participants) | 5
  Asian participants - [12C] Period 2 | 5.9 (4.5)
  Caucasian participants - [12C] Period 2: number analyzed (Participants) | 7
  Caucasian participants - [12C] Period 2 | 1.0 (1.2)

21. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: Up to Day 29 (MB Cohort) or up to Day 29 of Period 2 (AB Cohort)
Measure: Number; unit: Percentage of participants
Arm/Group | Absolute Bioavailability (BA) Cohort | Mass Balance (MB) Cohort
Number analyzed (Participants) | 16 | 6
Percentage of participants | 81.3 | 33.3

ADVERSE EVENTS:
Time Frame: MB Cohort: From Day -1 to Day 29 of Period 1 (approximately 30 days total). BA Cohort: from Day -1 of Period 1 up to Day 29 of Period 2 (approximately 60 days total).
Description: Safety data were analyzed by cohort rather than by period due to the well-established safety profile of RO7049389 from previous Phase 1 and Phase 2 studies. There was no difference in population in the BA cohort between Periods 1 and 2 and AEs were collected irrespective of intervention within the cohort.
Arm/Group | Absolute Bioavailability (BA) Cohort | Mass Balance (MB) Cohort
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6
Other Adverse Events (participants affected / at risk) | 13/16 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Absolute Bioavailability (BA) Cohort (N=16) | Mass Balance (MB) Cohort (N=6)
Eyelid rash (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 10 (10) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT04729309/Prot_SAP_000.pdf